CLINICAL TRIAL: NCT03798262
Title: Effect of Acute and Sub-acute Administration of Gluten on Extra-intestinal and Gastrointestinal Symptoms in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S58915
Record Dates: First submitted 2018-10-11; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteers, Gluten
MeSH Terms: interventions — Glutens

STUDY DESIGN:
Intervention Model Description: single-blinded, randomised controlled, cross-over study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten (Active Comparator): Patients receive 16 g of gluten acutely and afterwards 2 glutenfree muffins with 8 g of gluten for 5 days sub-acutely
  Interventions: Other: Gluten
- Placebo (Placebo Comparator): Patients receive 16 g of whey protein acutely and afterwards 2 glutenfree muffins for 5 days sub-acutely
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Gluten — Tereos
  Arms: Gluten
Other: Placebo — Whey protein from Nestlé Healthy Science
  Arms: Placebo

SUMMARY:
The investigators will investigate the effects of acute and sub-acute administration of gluten on mood, intestinal permeability, gastrointestinal symptoms and gut peptide levels in healthy volunteers (HV).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 20 - 25 kg/m2
* Stable body weight for at least 3 months prior to the start of the study

Exclusion Criteria:

* Medical

  * Coeliac disease (excluded either by absence of the HLA-DQ2 and HLA-DQ8 haplotype or by a normal duodenal biopsy (Marsh 0) performed at endoscopy while on a gluten containing diet in individuals expressing the HLA-DQ2 (human leukocyte antigen) or HLA-DQ8 haplotype)
  * Abdominal or thoracic surgery. Exception: appendectomy
  * Gastrointestinal, endocrine or neurological diseases
  * Cardiovascular, respiratory, renal or urinary diseases
  * Hypertension
  * Diagnosed food or drug allergies
* Psychiatric disorders
* Eating disorders
* Depressive disorders
* Anxiety disorders
* Psychotic disorders
* Restraint or emotional eating
* Dieters, especially no gluten-free diet or a diet low on gluten
* Medication on a regular basis, exception: oral contraception
* Smoking
* History of cannabis use or any other drug of abuse for at least 12 months prior to the study
* Alcohol abuse (more than 21 units of alcohol for men, more than 14 units for woman per week)
* Pregnant or breastfeeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
The effect of gluten acutely and sub-acutely on extraintestinal symptoms in HV measured on the Positive and Negative Affect Schedule | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 20), after test visit 3 (at day 36), after test visit 4 (at day 41)
  Change from baseline. Scores can be 'very slightly or not at all', 'a little', 'moderately', 'quite a bit', 'extremely'. Measured at day 0, day 15, day 20, day 36 and day 41.
The effect of gluten acutely and sub-acutely on extraintestinal symptoms in HV measured on the Profile of Mood State. | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 21), after test visit 3 (at day 36), after test visit 4 (at day 41)
  Change from baseline. Scores are measured on the Visual Analogue Scale. The scale is ranged 0 - 10, in which 0 no occurrence of the symptom and 10 a lot occurrence of the symptom. Measured at day 0, day 15, day 20, day 36 and day 41.

SECONDARY OUTCOMES:
The effect of gluten acutely and sub-acutely on gastrointestinal symptoms in HV measured on the visual analogue scale for gastrointestinal symptoms | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 21), after test visit 3 (at day 36), after test visit 4 (at day 41)
  Scores are measured on the Visual Analogue Scale. With '0' no complaints and '10' a lot of complaints (change from baseline).
The effect of gluten acutely and sub-acutely on intestinal permeability (using the lactulose mannitol ratio) | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 20), after test visit 3 (at day 36), after test visit 4 (at day 41)
  Investigate change in intestinal permeability after gluten administration. In the urine we can measure the ratio lactulose/mannitol. This can be measured using High Performance Liquid Chromatography
Effect of acute and sub-acute gluten administration on high sensitive reactive protein levels in blood samples | During test visit 0 (day 0), test visit 2 (at day 21), after test visit 4 (at day 41)
  Change in high sensitive reactive protein levels measured at day 0, day 21 and day 41.
Effect of acute and sub-acute gluten administration on Lipopolysaccharide-Binding Protein levels in blood samples | During test visit 0 (day 0), test visit 2 (at day 21), after test visit 4 (at day 41)
  Change in lipopolysaccharide-binding protein levels measured at day 0, day 21 and day 41.
Effect of acute and sub-acute gluten administration on Lipopolysaccharide levels in blood samples | During test visit 0 (day 0), test visit 2 (at day 21), after test visit 4 (at day 41)
  Change in lipopolysaccharide levels measured at day 0, day 21 and day 41.
Effect of acute and sub-acute gluten administration on gut microbiota composition (stool samples) | After test visit 0 (day 0), day 13 and day 14, after test visit 1 (day 15), day 16, 17, 18, 19 and 20, two days before test visit 3 (day 34 and 35), day 36, 37, 38, 39, 40
  Change in gut microbiota composition (compared to day 0) with focus on: Bifidobacterium, Lactobacillus, Enterobacteriaceae, E. coli; measured in stool samples. Analyses will provide an overall view of the gut microbiota composition.
Effect of acute and sub-acute gluten administration on cortisol awakening response (saliva samples) | Day before test visit 1 (day 14), test visit 1 (day 15), test visit 2 (day 21), day before test visit 3 (day 35), test visit 3 (day 36) and test visit 4 (day 41)
  Change in cortisol levels between gluten and placebo administration (saliva samples). Measured using an ELISA assay.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Jan Tack, Leuven
  - TARGID, Leuven

REFERENCES:
- [Derived] Iven J, Geeraerts A, Vanuytsel T, Tack J, Van Oudenhove L, Biesiekierski JR. Impact of Acute and Sub-Acute Gluten Exposure on Gastrointestinal Symptoms and Psychological Responses in Non-Coeliac Gluten Sensitivity: A Randomised Crossover Study. United European Gastroenterol J. 2025 Sep;13(7):1295-1306. doi: 10.1002/ueg2.70014. Epub 2025 Mar 26. PMID 40138597